CLINICAL TRIAL: NCT04116736
Title: ACUVUE® OASYS With Transitions™ Light Intelligent Technology™ Clinical Performance Registry
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-6334
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Vision Satisfaction in Bright Light

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- TEST Lens: Eligible subjects that are at least 18 years old, who have been recently fitted (within the last 2 months) with the ACUVUE® OASYS with Transitions™ will be asked to complete follow-up assessments performed online at approximately 2-weeks, 4-months, and 12-months following Visit 1.
  Interventions: Device: ACUVUE® OASYS with Transitions™
- CONTROL Lens: Eligible subjects that are at least 18 years old, who have been recently fitted (within the last 2 months) with spherical non-photochromic reusable marketed silicone hydrogel contact lenses (of any brand) will be asked to complete follow-up assessments performed online at approximately 2-weeks, 4-months, and 12-months following Visit 1.
  Interventions: Device: Silicone Hydrogel Contact Lens

INTERVENTIONS:
Device: ACUVUE® OASYS with Transitions™ — JJVC Marketed Contact Lens
  Other Names: TEST Lens
  Groups: TEST Lens
Device: Silicone Hydrogel Contact Lens — Any reusable spherical silicone hydrogel brand that is approved and marketed in the country conducting the study.
  Other Names: CONTROL Lens
  Groups: CONTROL Lens

SUMMARY:
This registry study is a one-year, one-visit, observational, prospective, open-label, two-arm, multi-center, multi-national, post-market study of approximately 300 patients who have recently been fitted with the ACUVUE® OASYS with Transitions™ and approximately 300 patients who have recently been fitted with spherical nonphotochromic reusable marketed silicone hydrogel contact lenses (of any brand). Eligible subjects will be asked to complete a Patient Registration Questionnaire several times throughout the year.

ELIGIBILITY:
Inclusion Criteria:

- Potential subjects must satisfy all of the following criteria to be enrolled in the study:

* Contact lens neophytes or those who have recently (i.e. within last 2 months) begun the use of a new lens type and have purchased a supply of lenses.
* A minimum age of 18 years, with no maximum age.
* The registrant must read and sign the Informed Consent form.
* The registrant must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

- Potential subjects who meet any of the following criteria will be excluded from participating in the study:

* Current participant in another research study.
* Employee or relative of site, or family member of Recruiting Practitioner or Johnson & Johnson.
* Non-spherical contact lens wearers, i.e. toric or multifocal lenses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be recruited from the clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials. Within the sites, subjects that have received a prescription of either Intervention within the last 2 months will be invited to participate without regard to any demographic or other ocular features.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (22):
- Spain (11):
  - Sanchez Rubal Ltd. - Sanchez Bregua, A Coruña
  - Sanchez Rubal Ltd - Finisterre, A Coruña
  - Optica Ronda, Almería
  - Natural Optics Balaguer, Balaguer
  - Centro Optico Raga, Linares
  - Centro Optico Montero, Madrid
  - Centro Boston de Optometria, Madrid
  - Cirugia Ocular de Madrid, Madrid
  - Opticalia Real Villa, Madrid
  - Opticas ClaraVision, Ontinyent
  - Centro Optico, Seville
- United Kingdom (11):
  - Eyesite Opticians, Reading, Berkshire
  - Leightons Insight Marlow, Marlow, Buckinghamshire
  - P Shah Opticians, London, England
  - Eyes On the Common Ltd., London, England
  - Hodd Barnes Dickens Ltd, London, England
  - Eyesite Opticians, Winchester, Hampshire
  - First Contact Opticians Ltd., Eastcote, Middlesex
  - Urquhart Opticians Ltd, Kilmarnock, Scotland
  - Eyesite Opticians, Weybridge, Surrey
  - Auckland Opticians, Horbury, Wakefield
  - Chalmers Opticians Ltd, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 146 subjects were enrolled in this study. All 146 subjects (88 in the Test group and 58 in the Control group) were deemed eligible at the screening visit. In the Control group 4 subjects were later identified as ineligible (enrolled in error), as they were wearing ineligible Control lenses. Of those enrolled, 113 subjects completed the study while 33 subjects were discontinued.
Groups:
- Test: Patients who had recently been fitted with ACUVUE® OASYS with Transitions™
- Control: Patients who had recently been fitted with spherical non-photochromic reusable marketed silicone hydrogel contact lenses of any brand.
Period: Overall Study
Arm/Group | Test | Control
Started | 88 | 58
Completed | 67 | 46
Not Completed | 21 | 12
Not completed — Withdrew consent during study | 3 | 1
Not completed — Subject no longer meets eligibility criteria | 1 | 4
Not completed — Subject withdrawn due to non-compliance to protocol | 11 | 7
Not completed — Switched to a different type of contact lens due to discomfort and dryness | 1 | 0
Not completed — Subject was enrolled in error | 2 | 0
Not completed — PI confirmed subject was not over 18 when enrolled in study. Subject discontinued | 1 | 0
Not completed — Subject did not like the lenses graduation change | 1 | 0
Not completed — Subject stopped wearing study lenses after 2 weeks due to dryness | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set including all enrolled subjects (signed consent form) regardless of subsequent withdrawal from study or deviation from protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 88 | 58 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (11.93) | 31.9 (12.09) | 33.1 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 40 | 91
  Male | 37 | 18 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Spain | 64 | 50 | 114
  United Kingdom | 24 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Vision Satisfaction in Bright Lighting - 2-Week Questionnaire
Description: Subjects will be asked to evaluate their vision satisfaction in bright lighting by rating their level of agreement with the statement "I am satisfied with the quality of my vision in bright lighting with these contact lenses" using a 5-point agreement Likert scale (Strongly Disagree, Disagree, Neither Agree Nor Disagree, Agree, and Strongly Agree). In the Control group 4 subjects were identified as ineligible after the screening visit because they were wearing ineligible Control lenses. Therefore, only 54 subjects were included in the Control group for the primary endpoint data summary. The number of missing responses in each lens group was reported.
Time Frame: 2-week questionnaire follow-up
Population: All subjects in the full analysis (FA) population excluding subjects that should have been deemed ineligible due to the new prescription of multifocal, toric, or daily disposable contact lenses at the screening visit. In the FA population, 4 out of 58 subjects were identified as ineligible after screening, resulting in 54 in the Control group among the analysis population. A summary of missing responses was reported for each endpoint at each timepoint.
Measure: Number; unit: Responses
Groups:
- Test: Subjects that wore the Test lens during the study.
- Control: Subjects that wore the Control lens during the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Strongly Agree | 33 | 21
  Agree | 33 | 24
  Neither Agree Nor Disagree | 10 | 2
  Disagree | 2 | 0
  Strongly Disagree | 0 | 0
  Missing Response (Subject didn't answer the item) | 10 | 7

2. Primary Outcome: Vision Satisfaction in Bright Lighting - 4-Month Questionnaire
Description: as for outcome 1
Time Frame: 4-month questionnaire follow-up
Population: as for outcome 1
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Strongly Agree | 24 | 20
  Agree | 38 | 25
  Neither Agree Nor Disagree | 7 | 2
  Disagree | 2 | 0
  Strongly Disagree | 0 | 0
  Missing Response (Subject didn't answer the item) | 17 | 7

3. Primary Outcome: Vision Satisfaction in Bright Lighting - 12-Month Questionnaire
Description: Subjects will be asked to evaluate their vision satisfaction in bright lighting by rating their level of agreement with the statement "I am satisfied with the quality of my vision in bright lighting with these contact lenses" using a 5-point agreement Likert scale (Strongly Disagree, Disagree, Neither Agree Nor Disagree, Agree, and Strongly Agree). In the Control group 4 subjects were identified as ineligible after the screening visit because they were wearing ineligible Control lenses. Therefore, only 54 subjects were included in the Control group for the primary endpoint data summary.
Time Frame: 12-month questionnaire follow-up
Population: as for outcome 1
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Strongly Agree | 23 | 22
  Agree | 29 | 21
  Neither Agree Nor Disagree | 4 | 2
  Disagree | 3 | 0
  Strongly Disagree | 0 | 0
  Missing Response (Subject didn't answer the item) | 29 | 9

4. Secondary Outcome: Overall Quality of Vision - 2-Week Questionnaire
Description: Overall quality of vision was assessed subjectively using the item "I am satisfied with the overall quality of my vision with these contact lenses". The item used a 5-point agreement scale: Strongly Disagree, Disagree, Neither Agree Nor Disagree, Agree, and Strongly Agree. In the Control group 4 subjects were identified as ineligible after the screening visit because they were wearing ineligible Control lenses. Therefore, only 54 subjects were included in the Control group for this secondary endpoint data summary. The number of missing responses in each lens group was reported.
Time Frame: 2-week questionnaire follow-up
Population: All subjects in the full analysis (FA) population excluding subjects that should have been deemed ineligible due to the new prescription of multifocal, toric, or daily disposable contact lenses at the screening visit. In the FA population, 4 out of 58 subjects were identified as ineligible after screening, resulting in 54 in the Control group among the analysis population. A summary of missing data was reported for each endpoint at each timepoint.
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Strongly Agree | 37 | 27
  Agree | 36 | 20
  Neither Agree Nor Disagree | 3 | 0
  Disagree | 1 | 0
  Strongly Disagree | 0 | 0
  Missing Response (Subject didn't answer the item) | 11 | 7

5. Secondary Outcome: Overall Quality of Vision - 4-Month Questionnaire
Description: as for outcome 4
Time Frame: 4-month questionnaire follow-up
Population: as for outcome 4
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Strongly Agree | 31 | 22
  Agree | 35 | 23
  Neither Agree Nor Disagree | 5 | 2
  Disagree | 0 | 0
  Strongly Disagree | 0 | 0
  Missing Response (Subject didn't answer the item) | 17 | 7

6. Secondary Outcome: Overall Quality of Vision - 12-Month Questionnaire
Description: as for outcome 4
Time Frame: 12-month questionnaire follow-up
Population: as for outcome 4
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Strongly Agree | 25 | 18
  Agree | 30 | 25
  Neither Agree Nor Disagree | 1 | 2
  Disagree | 3 | 0
  Strongly Disagree | 0 | 0
  Missing Response (Subject didn't answer the item) | 29 | 9

7. Secondary Outcome: Overall Comfort - 2-Week Questionnaire
Description: Overall comfort was assessed using the item "How would you rate the overall comfort of these contact lenses?". The item used the 5-point excellence scale, Excellent, Very Good, Good, Fair, and Poor. In the Control group 4 subjects were identified as ineligible after the screening visit because they were wearing ineligible Control lenses. Therefore, only 54 subjects were included in the Control group for this secondary endpoint data summary. The number of missing responses in each lens group was reported.
Time Frame: 2-week questionnaire follow-up
Population: as for outcome 4
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Excellent | 19 | 9
  Very Good | 37 | 28
  Good | 17 | 9
  Fair | 4 | 1
  Poor | 0 | 0
  Missing Response (Subject didn't answer the item) | 11 | 7

8. Secondary Outcome: Overall Comfort - 4-Month Questionnaire
Description: as for outcome 7
Time Frame: 4-month questionnaire follow-up
Population: as for outcome 4
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Excellent | 27 | 16
  Very Good | 25 | 19
  Good | 12 | 9
  Fair | 6 | 2
  Poor | 1 | 1
  Missing Response (Subject didn't answer the item) | 17 | 7

9. Secondary Outcome: Overall Comfort - 12-Month Questionnaire
Description: as for outcome 7
Time Frame: 12-month questionnaire follow-up
Population: as for outcome 4
Measure: Number; unit: Responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Responses
  Excellent | 20 | 10
  Very Good | 28 | 23
  Good | 8 | 9
  Fair | 2 | 2
  Poor | 1 | 1
  Missing Response (Subject didn't answer the item) | 29 | 9

10. Secondary Outcome: Pulfrich Effect
Description: Pulfrich effect was assessed subjectively using the item "While wearing these lenses, my depth perception of moving objects has NOT been impacted". Subjects who disagreed or strongly disagreed with the statement were considered to have experienced the Pulfrich effect. In the Control group 4 subjects were identified as ineligible after the screening visit because they were wearing ineligible Control lenses. Therefore, only 54 subjects were included in the Control group for this secondary endpoint data summary.
Time Frame: 2-week, 4-month, and 12-month questionnaire follow-up
Population: All subjects in the full analysis population excluding subjects that should have been deemed ineligible due to the new prescription of multifocal, toric, or daily disposable contact lenses at the screening visit. There were 58 subjects in Full Analysis population, but 4 subjects were identified as ineligible after the screening visit because they were wearing ineligible Control lenses. Therefore, only 54 subjects were included in the Control group for the secondary endpoint data summary.
Measure: Number; unit: Number of responses
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 54
Number of responses
  Number of Subjects Experienced the Pulfrich Effect at Least Once | 4 | 1
  Number of Subjects Experienced the Pulfrich Effect at 2-Week Evaluation | 4 | 0
  Number of Subjects Experienced the Pulfrich Effect at 4-Month Evaluation | 0 | 1
  Number of Subjects Experienced the Pulfrich Effect at 12-Month Evaluation | 0 | 0

11. Secondary Outcome: Serious or Significant Adverse Events
Description: A serious adverse event is any untoward medical occurrence that is potentially sight-threatening, requires hospitalization, results in persistent or significant disability / incapacity, or requires intervention to prevent permanent damage.
  Significant adverse events are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding serious adverse events).
Time Frame: Throughout the duration of the study, up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: Number of adverse events
Arm/Group | Test | Control
Number analyzed (Participants) | 88 | 58
Number of adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 12 months per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/58
Other Adverse Events (participants affected / at risk) | 0/88 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT04116736/Prot_SAP_000.pdf